CLINICAL TRIAL: NCT06674798
Title: School-based e-Health Non-Communicable Disease (NCD) Prevention Program to Improve Awareness in Adolescents From Urban Pakistan
Brief Title: School-based e-Health Non-Communicable Disease (NCD) Prevention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Fogarty International Center of the National Institutes of Health (Unknown)
Responsible Party: Principal Investigator, Dr Tazeen Saeed Ali, Professor, Aga Khan University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2023-9277-27367
Record Dates: First submitted 2024-10-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Noncommunicable Diseases; Health Knowledge, Attitudes, Practice; Non-communicable Disease Risk Factors
MeSH Terms: conditions — Noncommunicable Diseases; Behavior

STUDY DESIGN:
Intervention Model Description: Qualitative exploratory phase -quantitative intervention phase -qualitative explanatory phase
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, students will participate in 6 health promoting video sessions and three sessions will be delivered by trained facilitators per month. The session will be 30 to 40 minutes and the intervention will be provided over two months. The video material will be focused on the leading risk factors associated with NCDs as reported by different studies such as physical inactivity, unhealthy diet and overweight, obesity, harmful alcohol consumption and tobacco use.
  Interventions: Other: School-based eHealth NCD Prevention Program
- Control Group (No Intervention): The control group will not receive any intervention, and the end-line assessment will be conducted after two months of the intervention from both the groups. However, to maintain ethical standards, one session regarding NCDs and their associated risk factors will be delivered by trained facilitators to the control group after the end-line assessment.

INTERVENTIONS:
Other: School-based eHealth NCD Prevention Program — Students will participate in health-promoting sessions delivered by trained facilitators, with each session lasting 30 to 40 minutes. There will be a total of six health-promoting sessions conducted in the classroom for the intervention group, spanning two months with three sessions per month. The health-promoting videos from the school-based eHealth NCD prevention program will be shown in the classroom using multimedia. The drama-based videos will be developed in Urdu Language with English subtitles and will be based on based on contextually relevant content for the Pakistani secondary and higher secondary school students of age 13 to 18 years old. The content of these six sessions will be focused on the leading risk factors associated with NCDs as reported by different studies such as physical inactivity, unhealthy diet and overweight, obesity, harmful alcohol consumption and tobacco use.
  Arms: Intervention Group

SUMMARY:
The goal of this sequential mixed method study is to assess the feasibility and effectiveness of a school-based eHealth-NCD prevention program intervention to improve adolescents' knowledge, attitude, and practices regarding NCDs and associated risk factors. It aims :

1. To identify barriers and facilitators associated with implementing a school-based eHealth intervention to improve the knowledge, attitudes, and practices of secondary and higher secondary school students in Pakistan regarding NCDs and their associated risk factors.
2. To explore the stakeholders' perceptions regarding the design and content of the School based eHealth NCD prevention Program to improve the knowledge, attitudes, and practices of secondary and higher secondary school students in Pakistan regarding NCDs and their associated risk factors.
3. To assess the feasibility and effectiveness of the School-based eHealth NCD prevention program in secondary and higher secondary school in Karachi.
4. To evaluate the effectiveness of the school-based eHealth NCD prevention program in significantly improving the knowledge, attitudes, and practices of secondary and higher secondary school students in Karachi, Pakistan, regarding NCDs and their associated risk factors, as compared to a control group not receiving the intervention.
5. To explore the perceptions of students regarding the usefulness acceptability and task technology fit of the School-based eHealth NCD prevention Program in improving the knowledge, attitude, and practices of Pakistani Higher Secondary School students regarding NCDs and their associated risk factors.

Researcher aim to evaluate the effectiveness of the school-based eHealth NCD prevention program in significantly improving the knowledge, attitudes, and practices of secondary and higher secondary school students in Karachi, Pakistan, regarding NCDs and their associated risk factors, as compared to a control group not receiving the intervention.

Participants of intervention group will attend health-promoting sessions delivered by trained facilitators, with each session lasting 30 to 40 minutes. There will be a total of six health-promoting sessions be focused on the leading risk factors associated with NCDs as reported by different studies such as physical inactivity, unhealthy diet and overweight, obesity, harmful alcohol consumption and tobacco use will be conducted in the classroom for the intervention group.

DETAILED DESCRIPTION:
A sequential mixed methods design is used to allow a more robust exploration, validation, and explanation of the complex factors surrounding the implementation and effectiveness of a school-based eHealth NCD prevention program for currently enrolled grade 9-12 students in Karachi. The project progresses from initial exploration (qualitative exploration phase) to validation (quantitative phase) and deeper understanding (qualitative explanation phase), enhancing the study's overall rigor and validity. The qualitative exploration phase is based on an adaptation of the Technology Acceptance Model (TAM) and Task Technology Fit Model (TTFM).

Before starting the study, permission is obtained from the pertinent authorities at the provincial and district education departments, as well as from school principals. Consent will be sought from parents, while assent will be obtained from secondary and higher secondary school students. Scheduling of data collection will be coordinated with school administrators to ensure a suitable time. Trained data collectors will be responsible for gathering data on the school premises using interview-based questionnaires.

QUALITATIVE EXPLORATORY PHASE By starting with the exploratory qualitative phase, the study aims to explore the perceptions of secondary and higher secondary school students regarding the usefulness, acceptability, and task technology fitness of a school-based eHealth NCD prevention program in improving the knowledge, attitudes, and practices. A total of four FGDs (two groups of students and two groups of teachers) with eight participants each and at least ten key informant interviews (five from school administrators and five from parents) will be conducted. Consolidated Criteria for Reporting Qualitative Research (COREQ) guidelines will be used to analyze all qualitative data. The data will be audio-recorded, compiled, translated into English, and then analyzed using manual thematic analysis and Qualitative Solutions and Research International (QSR) NVivo version 10 for thematic-content analysis. All interviews and FGDs will be transcribed in English. Commonalities and differences across the data will be identified and clustered around thematic sections. Verbatim quotes will be added to complement the themes. This initial phase will yield rich contextual insights that can inform the design and content of the program.

QUANTITATIVE PHASE - INTERVENTION The subsequent quantitative phase will build upon the findings from the qualitative exploration phase, allowing for the systematic assessment of the program's feasibility and effectiveness in significantly improving the knowledge, attitudes, and practices of secondary and higher secondary school students in Karachi, Pakistan, regarding NCDs and their associated risk factors, as compared to a control group not receiving the intervention, using a clustered randomized controlled trial design. This sequential approach allows the researchers to utilize qualitative insights to inform the development of the quantitative phase, ensuring that the research process is informed and responsive to the complexities of the research context. The quantitative phase will then assess the feasibility and effectiveness of the intervention, validating and extending the qualitative findings.

With a desired statistical power of 0.8 and a confidence interval of 0.05, coupled with an anticipated effect size of 25%, the calculated sample size was found to be 247 participants. To account for potential attrition, a prudent approach involves adding a 10% attrition rate, resulting in a revised total sample size of 272 (136 individuals will be allocated to the intervention group and another 136 to the control group).

The randomization process for the allocation of the eight selected secondary and higher secondary schools in Karachi into either the intervention or control group will involve a clustered approach to enhance the robustness of the trial. The eight schools will be stratified based on their type (secondary or higher secondary) and gender (girls or boys), resulting in four strata. This ensures that the randomization process accounts for potential confounding variables associated with school type and gender.

Cluster Assignment: Each stratum, considered as a cluster, will be randomly assigned to either the intervention or control group. This helps minimize potential biases and enhances the internal validity of the study.

Randomization Sequence: A randomization sequence will be generated using a computer-based random number generator, specifying which clusters are allocated to the intervention and control groups.

Concealed Allocation: The allocation sequence will be concealed until the intervention begins, preventing selection bias. An independent researcher, not involved in the study implementation, will oversee the randomization process, enhancing transparency and minimizing the risk of systematic errors. This detailed clustered randomization strategy ensures that the intervention and control groups are balanced across important characteristics, allowing for a more accurate assessment of the impact of the school-based eHealth NCD prevention program on the knowledge, attitudes, and practices of Pakistani secondary and higher secondary school students while considering potential clustering effects within schools.

Due to the nature of the school-based eHealth NCD prevention program intervention, blinding of participants, instructors, and researchers is not feasible in this study.

After the random allocation of schools into intervention and control groups, baseline data regarding the awareness levels of students and students' weight and height will be measured (using calibrated weighing scales and stadiometers for accurate measurements) from both groups. Allocation will be revealed to the schools after recruitment and baseline assessment to avoid recruitment bias. Students in the intervention group will participate in health-promoting sessions delivered by trained facilitators. The health-promoting videos from the school-based eHealth NCD prevention program will be shown. The control group will not receive any intervention, and the end-line assessment will be conducted after two months of the intervention for both groups. However, to maintain ethical standards, one session regarding NCDs and their associated risk factors will be delivered by trained facilitators to the control group after the end-line assessment.

There will be six health-promoting video sessions in this segment. The audio of the videos will be in Urdu with English subtitles, and each video will be 8-12 minutes long. The sessions will be 30 to 40 minutes long, and the intervention will span two months with three sessions per month. The content of these six sessions will focus on the leading risk factors associated with NCDs, such as harmful alcohol consumption, tobacco use, physical inactivity, unhealthy diet, and overweight and obesity. The health education videos will be incorporated into classroom sessions using multimedia. Each session will consist of 25 to 35 students, with a trained facilitator guiding the discussions. Prior to implementing the intervention, a baseline qualitative assessment (adapted from the Global School Health Surveys, STEPwise Surveillance (STEPs) Survey of NCD risk factors, and a Mongolian survey questionnaire) will be conducted to explore the stakeholders' perceptions regarding the content and design of the web-based program. This pre-tested questionnaire will be available in both English and Urdu and will comprise three sections. The first section will contain sociodemographic information of the participants, the second section will contain questions about knowledge, attitudes, and practices related to NCDs (e.g., cardiovascular diseases, stroke, diabetes, hypertension), and the third section will cover questions on knowledge, attitudes, and practices related to NCDs' behavioral risk factors (e.g., diet, physical activity, and smoking). Based on these findings, the web-based program's content and design will be refined and modified as needed. The school-based eHealth program's conceptual framework, aimed at enhancing awareness of NCDs and associated risk factors, is rooted in the Theory of Planned Behavior (TPB)-that is, students' attitudes toward NCD prevention, societal expectations, and self-perceived control will shape their intentions and actions in adopting healthier habits. After the two-month intervention period, the same baseline questionnaire will be used to conduct a post-intervention survey among the participants, allowing for a comparison of their knowledge, attitudes, and practices before and after the program. This data will then be compared with the pre-assessment data to evaluate the impact of the intervention. The results will be presented in graphs and tables, offering visual representations of the participants' progress.

Data collected from respondents in this clustered randomized controlled trial (cRCT) will undergo a thorough analysis using appropriate methods to account for the clustered nature of the study design.

Descriptive analysis: Descriptive analysis will involve tabulating results as numbers (percentages) for qualitative variables and means (± standard deviation) for quantitative variables. To capture the cluster-level characteristics, summary statistics will be generated at both the individual and school levels.

Inferential analysis: Quantitative variables will be assessed for normality using the Shapiro-Wilk test. Given the clustered nature of the trial, a multilevel modeling approach, specifically linear mixed-effects models, will be employed to analyze quantitative outcomes. This approach is particularly suitable for accounting for within-cluster correlations. The analysis will include a comparison of baseline characteristics between the intervention and control groups. Appropriate statistical tests for categorical variables, such as chi-square tests, and continuous variables, such as independent t-tests or Mann-Whitney U tests based on distributional assumptions, will be utilized. To assess the effectiveness of the intervention, before-after data will be analyzed within each group using paired t-tests. Additionally, between-group analysis will be conducted using independent t-tests, comparing the change scores between the intervention and control groups.

Association analysis: Mixed-effects logistic regression models will be used to explore the associations between sociodemographic variables and changes in binary outcome variables (knowledge, attitude, and practice) while considering the clustering effect at the school level. Furthermore, mixed-effects linear regression models will be applied to assess the association of continuous outcome variables, such as knowledge scores and attitudes, with changes in self-reported practices. Random effects for schools will be explicitly specified to address the inherent clustering within the study design. Covariates for the multivariable analysis will be carefully chosen based on theoretical or empirical reasoning, avoiding the use of a stepwise approach to prevent overfitting and instability. Results from the analysis will be presented as adjusted odds ratios (OR) with corresponding 95% confidence intervals (CI). The significance level for all analyses will be set at 0.05, deeming any association with a p-value less than 0.05 as statistically significant.

QUALITATIVE -EXPLANATION Furthermore, the final qualitative explanatory phase will provide an in-depth understanding of students' perceptions regarding the usefulness, acceptability, and technological fitness of the program, adding depth and meaningful explanations to the quantitative findings. Two focus group discussions (FGDs) will be conducted with eight participants in each group. One FGD will be conducted with male students and one with female students.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (FGDs and Interviews)

* Students currently enrolled in secondary and higher secondary schools in Karachi and are in grades 9 to 12.
* Teachers who have been employed in secondary and higher secondary schools in Karachi for a minimum duration of 6 months.
* Parents or legal guardians of students who are currently enrolled in secondary and higher secondary schools in Karachi.
* Principals and vice principals of secondary and higher secondary schools in Karachi, District Education Officers, and decision-makers at Provincial Department of Education.

Phase 2 (Intervention)

- Both study and control group would be selected from secondary schools (students in grades 9-10) and Higher Secondary Schools (students in grades 11-12) located in Karachi, Pakistan

Phase 3 (FGDs) - Participants from grades 9 to 12 of the secondary and higher secondary schools who actively participated in the intervention and attended all the health-promoting sessions (equal representation of male and female)

Exclusion Criteria:

- Schools outside Karachi

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility (Recruitment rate) of the School-based eHealth NCD prevention program | 2 months
  Measurement Tool: Percentage of participants enrolled out of the total number invited.
  Units of Measure: Percentage (%). Description: It will be measured as the percentage of participants enrolled out of the total number of invited participants at baseline phase. The trial will be considered feasible if recruitment rates exceed 70%
To assess feasibility (Retention Rate) of the School-based eHealth NCD prevention program | 3 months
  Measurement Tool: Percentage of retained participants at 3 months among those initially recruited.
  Units of Measure: Percentage (%). Description: The retention rate will measure the percentage of participants who remain available for follow-up assessments at 3 months among those recruited initially. The trial will be considered feasible if retention rates exceed 70%
To assess feasibility (treatment fidelity) of the School-based eHealth NCD prevention program | 2 months
  Measurement Tool: Proportion of successfully conducted health-promoting sessions compared to planned sessions.
  Units of Measure: Proportion. Description: Treatment fidelity will be assessed as the proportion of health-promoting sessions that are successfully delivered as planned within the intervention period. A treatment fidelity rate above 70% will be used as a threshold for determining the program's feasibility in maintaining session integrity.
To assess effectiveness of the School-based eHealth NCD prevention program in improving the knowledge among secondary and higher secondary school students regarding the NCDs and their associated risk factors. | 2 months
  Measurement Tool: Knowledge will be assessed using a set of 26 questions adapted from study "An intervention program to reduce non-communicable diseases related behavioral risk factors among adolescents in institutional settings of Bangladesh".
  Units of Measure: Percentage score Description: Each question will be scored as either correct or incorrect, on the basis of standard medical textbooks and guidelines. The total knowledge score will be calculated, with a higher score indicating a better Knowledge. Based on previous Knowledge, Attitudes, and Practices (KAP) studies where a score of 60% or above has been used to categorize participants as having a satisfactory level of knowledge. This means that participants who achieve a score equal to or above 60% on the knowledge assessment will be considered to have a satisfactory level of knowledge regarding NCDs and their associated risk factors.
To assess effectiveness of the School-based eHealth NCD prevention program in improving the attitude among secondary and higher secondary school students regarding the NCDs and their associated risk factors. | 2 months
  Measurement Tool: A 14-item attitude questionnaire using a Likert scale adapted from study "An intervention program to reduce non-communicable diseases related behavioral risk factors among adolescents in institutional settings of Bangladesh"..
  Units of Measure: Total score of likert scale Description: Participants will be asked to rate each item on a 3-point scale, except for one item which will be rated on a 4-point scale. The scores will be added, and higher scores in the attitude section will indicate a more positive attitude towards NCDs' prevention. The attitude section will have a possible minimum score of 16 points and a possible maximum score of 49 points. In accordance with previous studies, the cut-off value for attitude will be set at 60%. This threshold is derived from existing research where a score of 60% or higher has been identified as an indicator of a positive or favorable attitude.
To assess effectiveness of the School-based eHealth NCD prevention program in improving the practices of secondary and higher secondary school students regarding the NCDs and their associated risk factors. | 2 months
  Measurement Tool: 22 questions will measure the dietary habits, physical activity, smoking, and substance abuse practices based on World Health Organization (WHO) recommendations and standard practices adapted from study "An intervention program to reduce non-communicable diseases related behavioral risk factors among adolescents in institutional settings of Bangladesh".
  1. Dietary risk behavior: presence of at least 2 of the 4 habits i.Inadequate fruit consumption: Less than 5 servings per day ii.Inadequate vegetable consumption: Less than 5 servings per day iii. Extra or raw salt consumption salt during every meal iv. Consuming Sugar Sweetened Beverage more than 3 days per week
  2. Physical Inactive: less than 60 min of physical activity of moderate intensity per day
  3. Smoking regularly in the last 30 days or exposed to passive smoking more than 3 days per week or any amount of alcohol intake or any substance abuse in the last 30 days will be regarded as at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tazeen Saeed Ali, Ph.D, Principal Investigator — Aga Khan University
Locations (7):
- Pakistan (7):
  - Allama Iqbal G.B.H.S.S FB Area, Karachi, Sindh
  - APWA G.G.H.S Liaquatabad, Karachi, Sindh
  - EAB G.G.S.S Block 6, Karachi, Sindh
  - G.B.H.S.S Farabi Muslimabad, Karachi, Sindh
  - G.G.H.S.S Gulshan e Iqbal Block 6, Karachi, Sindh
  - Junior Model School, Karachi, Sindh
  - Major Ziauddin School, Karachi, Sindh

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT06674798/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT06674798/ICF_001.pdf